CLINICAL TRIAL: NCT05416528
Title: Translation and Validation of the 8-item Contact Lens Dry Eye Questionnaire (CLDEQ-8) Among Chinese Soft Contact Lens Wearers
Brief Title: Chinese Translation and Validation of the 8-item Contact Lens Dry Eye Questionnaire (CLDEQ-8)
Acronym: CLDEQ-8
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao Yang, Professor Xiao Yang, M.D, PhD, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2022KYPJ100
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Contact Lens; Questionnaire; Contact Lens Discomfort
Keywords: the 8-item Contact Lens Dry Eye Questionnaire; CLDEQ-8; Contact Lens Discomfort; Questionnaire; Chinese translation and validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-cultural adaptation, evaluation and validation study of the 8-item Contact Lens Dry Eye Questionnaire (CLDEQ-8) among soft contact lens wearers in China.

DETAILED DESCRIPTION:
The aim of this study is to translate the 8-item Contact Lens Dry Eye Questionnaire (CLDEQ-8) into Chinese and evaluate its validity, and reliability among soft contact lens wearers in China. One hundred and thirty-four Chinese soft contact lens wearers will be included in the study. Subjects are required to complete the Chinese version of the 8-item Contact Lens Dry Eye Questionnaire (C-CLDEQ-8) on paper before eye examinations. A subgroup of 50 participants will be asked to complete C-CLDEQ-8 twice to evaluate the repeatability.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60
2. Native Chinese citizens with Chinese as first language
3. Wearing history with spherical disposable SCL (daily disposable, 2 weeks, or monthly disposable) for a least 1 months;
4. Willing to sign informed consent

Exclusion Criteria:

1. Any extended wear of SCLs, including wearing toric or multi-focal SCLs
2. Use SCL for monovision correction
3. Having clinically significant anterior segment abnormalities (including iritis and infection of the eye, lids, or ocular adnexa)
4. Having ocular or systemic disease that would preclude SCL wearing
5. Best corrected visual acuity of less than 0.8 in either eye
6. History of refractive or other types of corneal surgeries
7. Having eyelid abnormalities or functional ocular disorders that would induce relevant discomfort.

8) Having congenital or systemic conditions that would limit the capacity to answer the questionnaire

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects are residents of Guangzhou, China.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
The reliability of the C-CLDEQ-8 | before the ocular examination
  Subjects are asked to complete C-CLDEQ-8. Internal consistency (reliability) of the C-CLDEQ-8 is evaluated using the Cronbach's Alpha analysis and the corrected index of homogeneity. For Cronbach´s Alpha results: < 0.5 is considered unacceptable; 0.5-0.6 poor; 0.6-0.7 questionable; 0.7-0.8 acceptable; 0.8-0.9 good; and > 0.9 excellent.

SECONDARY OUTCOMES:
The repeatability of the C-CLDEQ-8 | before and after the ocular examination on the same day of visit
  a subgroup of 50 participants are asked to complete C-CLDEQ-8 twice. Intraclasss correlation coefficient between the two scores of the first and second questionnaire evaluation is used to evaluate the repeatability. >0.7 is considered reliable.
Cutoff score for C-CLDEQ-8 to predict "Excellent/Very Good" overall of SCLs. | before the ocular examination
  The Youden-index method is used to determine the cutoff value of the C-CLDEQ-8 score that maximized sensitivity+specificity -1.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China